CLINICAL TRIAL: NCT03413670
Title: Neural Mechanism Underlying Social Cognition in Depressive Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Normal University (Other)
Collaborators: Huilongguan Hospital (Unknown)
Responsible Party: Principal Investigator, ma, yina, Principal Investigator, Beijing Normal University
Other Study IDs: HLGdepression-fMRI
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the project, investigators plan to test difference of social cognition between depressive patients and healthy individuals and the brain activation underlying the difference to further understand the neural mechanism of depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 18 and 60
* Education experience above high school
* Score for Hamilton's Depression Scale >=17
* Diagnosis of depression through Scid

Exclusion Criteria:

* Undergoing electric shock treatment in 3 months
* Excluding those who with bipolar disorder
* Excluding those who with postpartum depression
* Excluding those who with hysteria

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Individuals diagnosed with depression and healthy control
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-02-08 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
emotion recognition | Baseline
  After viewing a video, participants will be asked to judge the person's attitude in the video. Through this paradigm, investigators could test emotional bias in social interaction in depressive patients.
resting state | Baseline
  In this part, investigators basically want to test the automatic neural activity for depressive patients while they are resting.
self-reflection | Baseline
  Participants will be asked to judge the discrepancy between actual self and ideal self.
response to negative stimuli | Baseline
  investigators used face-matching task to measure their response to negative stimuli. The participants will be asked to detect the identical face with same emotion.
structure | Baseline
  Investigators scanned structural images to detect the difference between clinical population and healthy population.
white matter | Baseline
  Investigators scanned DTI to detect the difference between clinical population and healthy population.

CONTACTS AND LOCATIONS:
Locations (1):
- Huilongguan Hospital, Beijing, China